CLINICAL TRIAL: NCT01537016
Title: WOUNDCHEK™ Protease Status Point of Care (POC) Diagnostic Test A Prospective, Multi Centre, Randomised, Clinical Study on Diabetic Foot Ulcers
Brief Title: WOUNDCHEK™ Protease Status Point of Care (POC) Diagnostic Test on DFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Systagenix Wound Management (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWM1215
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Promogran and High EPA (Experimental): Wound with high EPA will be treated with promogran and covered with a secondary dressing that is standard of care
  Interventions: Device: PROMOGRAN
- Promogran and Low EPA (Experimental): Wounds with low EPA will be treated with Promogran and covered with a secondary which is standard of care
  Interventions: Device: PROMOGRAN
- High EPA and standrad of care (Active Comparator): Wounds with high EPA will get standard of care as in line with current practice as they is no other test currently available for EPA
  Interventions: Device: Tielle
- Low EPA and standard of care (Active Comparator): Low EPA wounds will be treated with the standard of care for diabetic foot ulcers.
  Interventions: Device: Tielle

INTERVENTIONS:
Device: PROMOGRAN — PROMOGRAN® is a protease modulating dressing, formulated as a bioresorbable amorphous open-pored matrix constructed of 45% oxidised regenerated cellulose (ORC) and 55% bovine collagen
  Arms: Promogran and High EPA; Promogran and Low EPA
Device: Tielle — Tielle is a hydropolymer foam dressing that is designed to provide optimal wound healing
  Arms: High EPA and standrad of care; Low EPA and standard of care

SUMMARY:
The purpose of this trial is to determine if wounds with elevated protease activity (EPA) treated with targeted interventions such as protease modulating therapies can improve clinical and economic outcomes.

It is hypothesized that protease modulating dressings may provide significantly better clinical outcomes on EPA wounds over current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years old
* Patients with a diabetic foot ulcer as defined by Wagner grade 1 - 2
* ABPI of ≥0.6 to ensure ischemia will not impact healing
* No restriction on wound size or wound location
* Duration of ulcer ≥ 6 weeks ≤ 2 years
* The patient must be able to understand the trial and provide written informed consent
* No local or systemic signs of infection, with normal CRP and leukocyte levels below 10 000
* Wound has not been treated with PROMOGRAN® in 4 weeks prior to inclusion

Exclusion Criteria:

* Wound duration of less than 6 weeks or longer than 2 years
* Known hypersensitivity to any of the wound dressing used in the trial
* Current local or systemic antibiotics in the week prior to inclusion
* Patients with significant ischemia as defined by ABPI of ≤0.6
* Clinical infected wound as determined by the presence of 3 or more of the following clinical signs: perilesional erythema, pain between two dressing changes, malodorous wound, abundant exudate and oedema.
* Progressive neoplastic lesion treated by radiotherapy or chemotherapy
* Prolonged treatment with immunosuppressive agents or high dose corticosteroids
* Patients who have a current illness or condition which may interfere with wound healing in the last 30 days (carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse)
* Patients with renal insufficiency (with eGFR values <30 or on RRT) Life expectancy of <6 months
* Patients with uncontrolled diabetes as determined by Hb-A1c ≥ 12% ( = Hb-1CIFCC ≥ 107.65 mmol/mol)
* Patients who have participated in a clinical trial on wound healing within the past month
* Patients who are unable to understand the aims and objectives of the trial
* Patients with a known history of non adherence with medical treatment
* Females who are pregnant
* Subject has Acquired Immunodeficiency Syndrome (AIDS) or is known to be infected with Human Immunodeficiency Virus (HIV)
* Subject has viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
To identify EPA wounds using WOUNDCHEK™ Protease Status diagnostic test, and to compare the healing outcomes of two treatment regimes (PROMOGRAN®, a protease modulating therapy and current standard of care) on chronic wounds with EPA. | 4 weeks
  An improved healing outcome for diabetic foot ulcers ulcers will be defined as the proportion of wounds which reach a minimum 50% percentage reduction in wound surface area over a four-week treatment period.

SECONDARY OUTCOMES:
Reduction in wound area and cost effectiveness | 12 weeks
  The relative reductions in wound surface area from baseline over twelve weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, Prof, Principal Investigator — Cardiff University
Locations (5):
- Penn North Centers for advance wound care, Eire, Pennsylvania, United States
- Diabetes Klinik Bad Mergentheim Gmbh&CO. KG, Bad Mergentheim, Germany
- University of Pisa, Pisa, Italy
- Clinica Universitaria de Podologia, Madrid, Spain, Spain
- Bradford Royal Infirmary, Bradford, Yorkshire, United Kingdom